CLINICAL TRIAL: NCT03742466
Title: Local Injection of Ozone Versus Methylprednisolone Acetate in Carpal Tunnel Syndrome of Scleroderma Patients. A Single-blind Randomized Clinical Trial
Brief Title: Local Injection of Ozone Versus Methylprednisolone Acetate in Carpal Tunnel Syndrome of Scleroderma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Associate professor of Anesthesia, ICU, and pain, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17300356
Record Dates: First submitted 2018-11-10; First posted 2018-11-15 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Carpal Tunnel Syndrome; Chronic Pain; Scleroderma
MeSH Terms: conditions — Carpal Tunnel Syndrome; Chronic Pain; Scleroderma, Diffuse | interventions — Ozone; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone (Active Comparator): After prepping and draping the area, intracarpal injection of ozone/oxygen mixture (20 ml, 25μg/ml) will be performed under sonographic guidance
  Interventions: Drug: Ozone
- methylprednisolone acetate (Active Comparator): After prepping and draping the area, intracarpal injection of methylprednisolone acetate 40mg, and 40 mg lidocaine (20 ml, volume) will be performed under sonographic guidance
  Interventions: Drug: methylprednisolone acetate

INTERVENTIONS:
Drug: Ozone — After prepping and draping the area, intracarpal injection of ozone/oxygen mixture (20 ml, 25μg/ml) will be performed under sonographic guidance
  Arms: Ozone
Drug: methylprednisolone acetate — After prepping and draping the area, intracarpal injection of methylprednisolone acetate 40mg, and 40 mg lidocaine (20 ml, volume) will be performed under sonographic guidance
  Arms: methylprednisolone acetate

SUMMARY:
Carpal tunnel syndrome is a common peripheral entrapment neuropathy, this study aims to investigate if, and to what extent local ozone therapy could offer symptom improvement in scleroderma patients with Carpal tunnel syndrome

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression syndrome the upper extremities. Its problem has a high prevalence ranged estimated prevalence of 3.8% in the general population, 3 and 7.8% in the working population. It occurs at any age, especially in individuals in their 40s to 60s, and the male: female ratio is reported to be 3:7. A lot of treatment modalities have been tried to improve the condition, starting from local anesthetic injection, steroid, and up to surgical decompression of the nerves.

Scleroderma patients are a special group which usually sufferers from such problem

ELIGIBILITY:
Inclusion Criteria:

* adult patients with scleroderma
* complaining of carpal tunnel syndrome of 3-month duration or more
* diagnosed axonal neuropathy using electrodiagnosis, nerve conduction study

Exclusion Criteria:

* patient refusal
* infection at the site of intervention
* previous injection in the recent 3 months
* Coagulopathy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
to assess pain alleviation through the visual analog scale (VAS) | 6 months
  visual analog scale of pain value of (0 cm) no pain , and value of (10 cm) worst pain

SECONDARY OUTCOMES:
Changes in median nerve conduction parameters | 6 months
  distal motor latency

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No